CLINICAL TRIAL: NCT03842189
Title: A Multicenter, Open-label Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of M281 Administered to Pregnant Women at High Risk for Early Onset Severe Hemolytic Disease of the Fetus and Newborn (HDFN)
Brief Title: A Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of M281 Administered to Pregnant Women at High Risk for Early Onset Severe Hemolytic Disease of the Fetus and Newborn (HDFN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108980; MOM-M281-003 (Other: Janssen Research & Development, LLC); 2017-004958-42 (EudraCT Number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hemolytic Disease of the Fetus and Newborn
Keywords: M281; Hemolytic Disease of the Fetus and Newborn; HDFN; Rhesus Disease; Hemolytic disease due to fetomaternal alloimmunization; Hemolytic disease of the newborn with Kell alloimmunization; Rhesus (Rh) isoimmunization of foetus or newborn; Isoimmunization due to other red cell factors; ABO isoimmunization of foetus or newborn; Haemolytic anaemia due to other unclassified antibodies; Isoimmune; Isoimmunized; Isoimmunization; Alloimmune; Alloimmunized; Alloimmunization; Pregnant women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M281 (Experimental)
  Interventions: Drug: M281

INTERVENTIONS:
Drug: M281 — Participants will receive once weekly intravenous (IV) infusions of M281

SUMMARY:
The purpose of this study is to evaluate the safety in mother and neonate/infant of M281 administered to pregnant women who are at high risk for Early Onset Severe Hemolytic Disease of the Fetus and Newborn (EOS-HDFN). The effectiveness of the investigational drug M281 will be measured by looking at the percentage of participants with live birth at or after gestational age (GA) 32 weeks and without a need for an intrauterine transfusion (IUT) throughout their entire pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Approximately 15 eligible participants and their offspring will be enrolled
* Each participant must meet all of the following criteria to be enrolled in the study:
* Female and greater than or equal to (>=)18 years of age
* Pregnant to an estimated gestational age of between 8 up to 14 weeks
* A previous pregnancy with a gestation that included at least one of the following prior to week 24 gestation:
* Severe fetal anemia, defined as hemoglobin less than or equal to (<=) 0.55 multiples of the median (MOM) for gestational age
* Fetal hydrops with peak systolic velocity MOM >=1.5
* Stillbirth with fetal or placental pathology indicative of hemolytic disease of the fetus and newborn (HDFN)
* Maternal alloantibody titers for anti-D of >=32, or anti-Kell titers >=4
* Free fetal deoxyribonucleic acid consistent with an antigen-positive fetus (blood sample taken from mother)
* Maternal evidence for Immunity to measles mumps, rubella, and varicella, as documented by serologies performed during Screening. If initial serologies are borderline or negative, they may be repeated at a second lab. Alternatively, vaccination records can be used to support evidence of immunity.
* Screening immunoglobulin G and albumin levels within the laboratory normal range for gestational age of pregnancy
* Willing to receive standard of care with intrauterine transfusion if clinically indicated
* Agree to receive recommended vaccinations per local standard of care for both mother and child throughout the course of the study
* It is recommended that patients are up-to-date on age-appropriate vaccinations prior to screening as per routine local medical guidelines. For study patients who received locally-approved (and including emergency use-authorized) Coronavirus Disease 2019 (COVID-19) vaccines recently prior to study entry, follow applicable local vaccine labelling, guidelines, and standard of care for pregnant women receiving immune-targeted therapy when determining an appropriate interval between vaccination and study enrollment

Exclusion Criteria:

* Currently pregnant with multiples (twins or more)
* Pre-eclampsia In current pregnancy or history of pre-eclampsia in a previous pregnancy
* Gestational hypertension in the current pregnancy
* Current unstable hypertension
* History of severe or recurrent pyelonephritis, 4 or more lower urinary tract infections in the past year or in a previous pregnancy
* History of genital herpes infection
* Active Infection at Screening or Baseline with Coxsackie, syphilis, cytomegalovirus, toxoplasmosis or herpes simplex 1 or 2, as evidenced by clinical signs and symptoms (evidence for prior Infection or exposure, but without clinical signs and symptoms of active infection is acceptable)
* Active infection with tuberculosis as evidenced by positive QuantiFERON-tuberculosis testing
* Requires treatment with corticosteroids or immunosuppression for disorders unrelated to the pregnancy (use of low-potency topical corticosteroids or intra-articular corticosteroids is permitted)
* Has received or is expected to receive any live virus or bacterial vaccine within 12 weeks prior to screening or has a known need to receive a live vaccine while receiving nipocalimab, or within 12 weeks after the last administration of nipocalimab in the study or has received Bacille Calmett-Guérin (BCG) vaccine within 1 year prior to the first administration of nipocalimab
* Currently receiving an antibody-based drug or an Fc-fusion protein drug
* Received plasmapheresis and/or intravenous immunoglobulin during the current pregnancy for treatment of HDFN
* COVID-19 infection: during the 6 weeks prior to baseline (regardless of vaccination status), have had any of: a) confirmed severe acute respiratory syndrome coronavirus(-2) (SARS-CoV-2) (COVID-19) infection (test positive), or; b) suspected SARS-CoV-2 infection (clinical features without documented test results), or; c) close contact with a person with known or suspected SARS-CoV-2 infection. Exception: may be included with a documented negative result for a validated SARSCoV-2 test: obtained at least 2 weeks after conditions a), b), c) above (timed from resolution of key clinical features if present, example fever, cough, dyspnea) and; with absence of all conditions a), b), c) above during the period between the negative test result and the baseline study visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Liverpool Hospital, Sydney, Australia
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUM - Centre hospitalier universitaire de Montreal, Montreal, Quebec
- Justus-Liebig-Universität Gießen, Kinderherzzentrum, Giessen, Germany
- Leiden University Medical Center, Leiden, Netherlands
- Hosp. Univ. San Cecilio, Granada, Spain
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - University College London Hospitals NHSFT, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Winter DP, Moise KJ, Ling LE, Oepkes D, Tiblad E, Joanne Verweij EJT, Smoleniec J, Sachs UJ, Bein G, Kilby MD, Miller RS, Devlieger R, Streisand JB, Bredius RGM, Cafone J, Lam E, Leu JH, Mirza A, Nelson RM, Smith V, Schwartz LB, Tjoa ML, Saeed-Khawaja S, Komatsu Y, Lopriore E. Infant Immunity after Maternal Nipocalimab in Severe Hemolytic Disease of the Fetus and Newborn. NEJM Evid. 2026 Feb;5(2):EVIDoa2500097. doi: 10.1056/EVIDoa2500097. Epub 2026 Jan 27. PMID 41591368
- [Derived] Moise KJ Jr, Ling LE, Oepkes D, Tiblad E, Verweij EJTJ, Lopriore E, Smoleniec J, Sachs UJ, Bein G, Kilby MD, Miller RS, Devlieger R, Audibert F, Emery SP, Markham K, Norton ME, Ocon-Hernandez O, Pandya P, Pereira L, Silver RM, Windrim R, Streisand JB, Leu JH, Mirza A, Smith V, Schwartz LB, Tjoa ML, Saeed-Khawaja S, Komatsu Y, Bussel JB; UNITY Study Group. Nipocalimab in Early-Onset Severe Hemolytic Disease of the Fetus and Newborn. N Engl J Med. 2024 Aug 8;391(6):526-537. doi: 10.1056/NEJMoa2314466. PMID 39115062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled population included 13 maternal participants and 12 neonates born to maternal participants. There was one stillbirth which was not considered enrolled. Only livebirths were included in analyses and presented below.
Pre-assignment Details: Initial drug dose was 30 milligrams per kilogram(mg/kg) based on baseline weight (BLW). Per protocol amendments, dose increased to 45 mg/kg BLW, later adjusted to 45 mg/kg based on time-adjusted weight (weight at most recent biweekly visit) to allow dosing interval without loss of receptor occupancy to account for weight increases during pregnancy.
Groups:
- Group 1 (Maternal): 30 mg/kg BLW: Maternal participants received a single dose intravenous (IV) infusion of nipocalimab 30 milligrams per kilograms (mg/kg) based on baseline weight (BLW), once weekly from gestation age (GA) Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [Postpartum {PP} Week 24]).
- Group 2 (Maternal): 30 to 45 mg/kg BLW: Maternal participants received a single dose IV infusion of nipocalimab 30 mg/kg initially based on BLW followed by nipocalimab 45 mg/kg with increase in weight, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 3 (Maternal): 45 mg/kg BLW: Maternal participants received a single dose IV infusion of nipocalimab 45 mg/kg based on BLW, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 4 (Maternal): 45 mg/kg TAW: Maternal participants received a single dose IV infusion of nipocalimab 45 mg/kg based on time-adjusted weight (TAW), once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 1 (Neonates and Infants): 30 mg/kg BLW: Neonates and infants born to mothers from Group 1 were followed up for safety from postpartum (PP) Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
- Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW: Neonates and infants born to mothers from Group 2 were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
- Group 3 (Neonates and Infants): 45 mg/kg BLW: Neonates and infants born to mothers from Group 3 were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
- Group 4 (Neonates and Infants): 45 mg/kg TAW: Neonates and infants born to mothers from Group 4 were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
Period: Overall Study
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW
Started | 3 | 2 | 4 | 4 | 3 | 2 | 4 | 3
Completed | 3 | 2 | 4 | 4 | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | Total
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 3 | 2 | 4 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The total column presents the mean and standard deviation for only maternal participants.
  Years | 38.7 (1.53) | 37.0 (1.41) | 38.3 (4.43) | 30.8 (4.19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 35.8 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 4 | 3 | 1 | 0 | 0 | 17
  Male | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 4 | 4 | 3 | 2 | 3 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
    Not Hispanic or Latino | 2 | 2 | 4 | 4 | 2 | 2 | 4 | 3 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 5
  Belgium | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Germany | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 4
  Netherlands | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4
  Sweden | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4
  United Kingdom | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  United States | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Maternal Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TEAE was defined as any event occurring after the initiation of the first infusion of nipocalimab.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to Postpartum (PP) Week 24 (up to 50 weeks)
Population: Safety analysis set included all maternal participants who had received at least 1 dose of nipocalimab.
Measure: Count of Participants; unit: Participants
Groups:
- Group 4 (Maternal): 45 mg/kgTAW: Maternal participants received a single dose IV infusion of nipocalimab 45 mg/kg based on time-adjusted weight (TAW), once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow-up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- All Maternal Participants: Maternal participants of Group 1 (30 mg/kg BLW), Group 2 (30 to 45 mg/kg BLW), Group 3 (45 mg/kg BLW), and Group 4 (45 mg/kg TAW) who received a single dose of IV infusions of nipocalimab once weekly from gestation age (GA) Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Participants | 3 | 2 | 4 | 4 | 13

2. Primary Outcome: Number of Neonates/Infants With Adverse Events (AEs)
Description: An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Time Frame: From Birth (PP Day 0) up to PP Week 96
Population: Neonates or infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy.
Measure: Count of Participants; unit: Participants
Groups:
- All Neonates and Infants: All neonates and infants born to mothers from Group 1 (30 mg/kg BLW), Group 2 (30 to 45 mg/kg BLW), Group 3 (45 mg/kg BLW), and Group 4 (45 mg/kg TAW) were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants | 3 | 2 | 4 | 3 | 12

3. Primary Outcome: Number of Maternal Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: SAE was defined as any untoward medical occurrence that resulted in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TESAEs were any SAEs occurring after the initiation of the first infusion of nipocalimab.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to PP Week 24 (up to 50 weeks)
Population: Safety analysis set included all maternal participants who had received at least 1 dose of nipocalimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Participants | 2 | 0 | 1 | 2 | 5

4. Primary Outcome: Number of Neonates/Infants With Serious Adverse Events (SAEs)
Description: SAE was defined as any untoward medical occurrence that resulted in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Time Frame: From Birth (PP Day 0) up to PP Week 96
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 (Neonates and Infants): 30 mg/kg BLW: Neonates and infants born to mothers from Group 1 were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any nipocalimab study drug.
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants | 2 | 1 | 1 | 2 | 6

5. Primary Outcome: Number of Maternal Participants With Treatment-emergent Adverse Events of Special Interest (TEAESIs)
Description: Number of maternal participants with TEAESIs were reported. An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. All infections requiring anti-infective (that is, oral or intravenous antibacterial, antiviral, or antifungal) treatment and with hypoalbuminemia greater than or equal to (>=) Grade 3 (less than [<]20 gram per liter [g/L] by National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 criteria were considered an AESI for maternal participants. TEAE was defined as any event occurring after the initiation of the first infusion of nipocalimab.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to PP Week 24 (up to 50 weeks)
Population: Safety analysis set included all maternal participants who had received at least 1 dose of nipocalimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Participants
  Infections: Treatment with Oral /Intravenous | 1 | 1 | 1 | 2 | 5
  Hypoalbuminemia <20 g/L | 0 | 0 | 0 | 0 | 0
  Overall AESIs | 1 | 1 | 1 | 2 | 5

6. Primary Outcome: Number of Neonates/Infants With Adverse Events of Special Interest (AESIs)
Description: Number of neonates/infants with TEAESIs were reported. An AE was any unfavorable and unintended sign (example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. All infections requiring anti-infective (that is, oral or intravenous antibacterial, antiviral, or antifungal) treatment, unexpected/unusual childhood illnesses and Immunoglobulin G (IgG) concentrations <200 milligrams per deciliter (mg/dL) at Week 24 through Week 47 or <300 mg/dL at Week 48 through Week 96 were considered an AESI for neonates and infants.
Time Frame: From birth (PP Day 0) up to PP Week 96
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- All Neonates and Infants: All neonates and infants born to mothers from Group 1 (30 mg/kg BLW), Group 2 (30 to 45 mg/kg BLW), Group 3 (45 mg/kg BLW), and Group 4 (45 mg/kg TAW) were followed up for safety from PP Day 0 up to 96 weeks. Neonates and infants in this group did not receive any study drug.
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants
  IgG Concentrations <200 mg/dL | 1 | 2 | 0 | 0 | 3
  Infections: Treatment with Oral /Intravenous | 0 | 1 | 0 | 1 | 2
  Unexpected/Unusual Childhood Illnesses | 0 | 0 | 0 | 0 | 0
  Overall AESI | 1 | 2 | 0 | 1 | 4

7. Primary Outcome: Maternal Participants: Absolute Value of Electrocardiogram (ECG) Parameter - Mean Ventricular Rate at Baseline
Description: Absolute value of ECG parameter - mean ventricular rate at baseline in maternal participants was reported. Electrocardiogram assessments included comments on whether the tracings were normal or abnormal, rhythm, presence of arrhythmia or conduction defects, morphology, any evidence of myocardial infarction, or ST segment, T Wave, and U Wave abnormalities.
Time Frame: Baseline (GA Week 14)
Population: The full analysis set (FAS) included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Beats per minute | 77.0 (10.58) | 77.5 (3.54) | 63.0 (5.35) | 76.3 (8.42) | 72.5 (9.41)

8. Primary Outcome: Maternal Participants: Absolute Value of Electrocardiogram (ECG) Parameter - Mean Ventricular Rate at GA Week 36
Description: Absolute value of ECG parameter - mean ventricular rate at GA Week 36 in maternal participants was reported. Electrocardiogram assessments included comments on whether the tracings were normal or abnormal, rhythm, presence of arrhythmia or conduction defects, morphology, any evidence of myocardial infarction, or ST segment, T Wave, and U Wave abnormalities.
Time Frame: GA Week 36
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Beats per minute | 89.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 77.0 (21.21) | 80.7 (7.51) | 77.0 (21.21) | 79.9 (12.71)

9. Primary Outcome: Maternal Participants: Change From Baseline in ECG Parameter- Mean Ventricular Rate
Description: Change from baseline in ECG parameter- mean ventricular rate in maternal participants was reported. Electrocardiogram assessments included comments on whether the tracings were normal or abnormal, rhythm, presence of arrhythmia or conduction defects, morphology, any evidence of myocardial infarction, or ST segment, T Wave, and U Wave abnormalities.
Time Frame: Baseline (GA Week 14) and GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Beats per minute | 8.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -0.5 (24.75) | 16.7 (7.37) | 8.0 (22.63) | 9.1 (15.08)

10. Primary Outcome: Number of Maternal Participants With Treatment-emergent (TE) Clinically Important Laboratory and Biomarker Immunoglobulin G (IgG) Values Over Time
Description: Laboratory parameters included hematology, chemistry, blood Lipids panel, and Immunoglobulin G (IgG) parameters. TEAE was defined as any event occurring after the initiation of the first infusion of nipocalimab. Here, HDL: high-density lipoprotein, LDL: low-density lipoprotein. The during-pregnancy value of albumin <20 g/L was from a local laboratory and was >=20 g/L when analyzed at the central laboratory for the same time point.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to PP Week 24 (up to 50 weeks)
Population: The safety analysis set included all maternal participants who had received at least 1 dose of nipocalimab. Here, n (number analyzed): number of participants evaluable for each category. n=0 signifies no participant was available for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Participants
  During pregnancy: Cholesterol >9.025 millimoles per liter (mmol/L) | 1 | 2 | 3 | 2 | 8
  During pregnancy: LDL >5.793 mmol/L: number analyzed (Participants) | 0 | 1 | 2 | 4 | 7
  During pregnancy: LDL >5.793 mmol/L |  | 0 | 1 | 2 | 3
  During pregnancy: HDL Cholesterol <1.2413 mmol/L: number analyzed (Participants) | 0 | 1 | 2 | 4 | 7
  During pregnancy: HDL Cholesterol <1.2413 mmol/L |  | 0 | 0 | 0 | 0
  During pregnancy: Triglycerides >5.114 mmol/L | 0 | 0 | 1 | 1 | 2
  During pregnancy: Albumin <20 grams per Liter (g/L) | 0 | 0 | 0 | 1 | 1
  During pregnancy: Immunoglobulin G <1 g/L | 1 | 0 | 1 | 0 | 2
  Post Birth: Cholesterol >5.172 mmol/L | 3 | 2 | 4 | 2 | 11
  Post Birth: LDL >2.586 mmol/L: number analyzed (Participants) | 0 | 1 | 2 | 4 | 7
  Post Birth: LDL >2.586 mmol/L |  | 1 | 2 | 3 | 6
  Post Birth: HDL <1.0344 mmol/L: number analyzed (Participants) | 0 | 1 | 2 | 4 | 7
  Post Birth: HDL <1.0344 mmol/L |  | 0 | 1 | 0 | 1
  Post Birth: Triglycerides >1.6935 mmol/L | 1 | 1 | 3 | 2 | 7
  Post Birth: Albumin <20 g/L | 0 | 0 | 0 | 0 | 0
  Post Birth: Immunoglobulin G <1 g/L | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Neonates or Infants With Clinically Important Laboratory and Biomarker Immunoglobulin G (IgG) Values Over Time
Description: Laboratory parameters included total bilirubin and biomarker included immunoglobulin G (IgG).
Time Frame: From Birth (PP Day 0) up to PP Week 96
Population: The neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Only those categories in which at least one neonates or Infants had data were reported in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants
  Total Bilirubin >136.8 mmol/L | 1 | 1 | 3 | 3 | 8
  Immunoglobulin G < 1 g/L | 1 | 0 | 0 | 0 | 1
  Immunoglobulin G < 2 g/L | 2 | 2 | 4 | 2 | 10

12. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Temperature at Baseline
Description: Absolute value of vital signs - body temperature at baseline in maternal participants was reported.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Degree Celsius | 36.6 (0.1) | 37.0 (0.5) | 37.2 (0.5) | 36.8 (0.8) | 36.9 (0.6)

13. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Temperature at GA Week 36
Description: Absolute value of vital signs - body temperature at GA Week 36 in maternal participants was reported.
Time Frame: GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
Degree Celsius | 36.7 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 36.8 (0.0) | 37.1 (0.5) | 36.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 36.8 (0.5)

14. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Temperature at PP Week 24
Description: Absolute value of vital signs - body temperature at PP Week 24 in maternal participants was reported.
Time Frame: PP Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Degree Celsius | 36.5 (0.1) | 36.8 (0.3) | 36.8 (0.3) | 36.7 (0.5) | 36.7 (0.3)

15. Primary Outcome: Maternal Participants: Change From Baseline in Vital Sign - Body Temperature
Description: Change from baseline in vital signs- body temperature in maternal participants was reported.
Time Frame: Baseline (GA Week 14), GA Week 36, and PP Week 24
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and n (number analyzed) signifies number of participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Degree Celsius
  GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
  GA Week 36 | 0.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -0.2 (0.5) | -0.2 (0.0) | 0.2 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -0.1 (0.3)
  PP Week 24 | -0.1 (0.1) | -0.2 (0.2) | -0.5 (0.7) | -0.1 (1.0) | -0.2 (0.7)

16. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Respiratory Rate at Baseline
Description: Absolute value of vital signs -respiratory rate at baseline in maternal participants was reported.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
breaths per minute | 17.0 (1.7) | 19.0 (1.4) | 15.5 (3.4) | 18.0 (2.8) | 17.2 (2.7)

17. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Respiratory Rate at GA Week 36
Description: Absolute value of vital signs -respiratory rate at GA Week 36 in maternal participants was reported.
Time Frame: GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
Breaths per minute | 20.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 18.0 (0.0) | 16.3 (3.2) | 17.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 17.4 (2.3)

18. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Respiratory Rate at PP Week 24
Description: Absolute value of vital signs - respiratory rate at PP Week 24 in maternal participants was reported.
Time Frame: PP Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Breaths per minute | 16.5 (2.1) | 15.5 (2.1) | 15.8 (3.9) | 17.3 (3.6) | 16.3 (3.0)

19. Primary Outcome: Maternal Participants: Change From Baseline in Vital Sign - Respiratory Rate
Description: Change from baseline in vital signs- respiratory rate in maternal participants was reported.
Time Frame: Baseline (GA Week 14), GA Week 36, and PP Week 24
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, n (number analyzed) signifies number of participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Breaths per minute
  GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
  GA Week 36 | 2.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -1.0 (1.4) | 1.0 (1.0) | 1.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.6 (1.4)
  PP Week 24 | 0.0 (0.0) | -3.5 (0.7) | 0.3 (1.3) | -0.8 (3.0) | -0.8 (2.2)

20. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Pulse Rate at Baseline
Description: Absolute value of vital signs - pulse rate at baseline in maternal participants was reported.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Beats per minute | 81.3 (8.7) | 81.0 (8.5) | 67.5 (4.2) | 73.5 (8.9) | 74.6 (8.8)

21. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Pulse Rate at GA Week 36
Description: Absolute value of vital signs -pulse rate at GA Week 36 in maternal participants was reported.
Time Frame: GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
beats per minute | 88.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 95.0 (17.0) | 84.0 (9.5) | 100.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 90.0 (11.0)

22. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs -Pulse Rate at PP Week 24
Description: Absolute value of vital signs -pulse rate at PP Week 24 in maternal participants was reported.
Time Frame: PP Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Beats per minute | 73.0 (2.8) | 75.0 (4.2) | 69.8 (10.2) | 77.8 (4.1) | 73.8 (6.9)

23. Primary Outcome: Maternal Participants: Change From Baseline in Vital Sign - Pulse Rate
Description: Change from baseline in vital signs -pulse rate in maternal participants was reported.
Time Frame: Baseline (GA Week 14), GA Week 36, and PP Week 24
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Beats per minute
  GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 1 | 7
  GA Week 36 | -3.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 14.0 (8.5) | 15.0 (6.1) | 29.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 14.1 (10.5)
  PP Week 24 | -3.5 (6.4) | -6.0 (4.2) | 2.3 (8.5) | 4.3 (11.4) | 0.6 (8.8)

24. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Baseline
Description: Absolute value of vital signs - SBP and DBP at baseline in maternal participants was reported.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Millimeter of mercury
  SBP | 112.0 (11.3) | 100.5 (3.5) | 102.3 (4.6) | 104.8 (12.4) | 105.0 (9.2)
  DBP | 68.7 (3.5) | 59.5 (3.5) | 63.3 (6.9) | 64.5 (10.8) | 64.3 (7.3)

25. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at GA Week 36
Description: Absolute value of vital signs -SBP and DBP at GA Week 36 in maternal participants was reported.
Time Frame: GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Millimeter of mercury (mmHg)
  SBP | 134.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 105.0 (8.5) | 107.3 (9.6) | 110.5 (7.8) | 110.9 (11.7)
  DBP | 70.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 73.0 (5.7) | 66.3 (4.2) | 69.0 (5.7) | 69.1 (4.7)

26. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at PP Week 24
Description: Absolute value of vital signs - SBP and DBP at PP Week 24 in maternal participants was reported.
Time Frame: PP Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Millimeters of mercury
  SBP | 117.5 (14.8) | 110.5 (14.8) | 112.3 (4.0) | 118.8 (9.9) | 115.0 (9.2)
  DBP | 73.5 (10.6) | 69.5 (6.4) | 71.3 (6.2) | 71.8 (1.7) | 71.5 (5.2)

27. Primary Outcome: Maternal Participants: Change From Baseline in Vital Sign - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline in vital signs -SBP and DBP in maternal participants were reported.
Time Frame: Baseline (GA Week 14), GA Week 36, and PP Week 24
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and n (number analyzed): number of participants evaluable for specified categories and timepoints.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Millimeters of mercury
  SBP: GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
  SBP: GA Week 36 | 15.0 (NA) — "NA signifies that SD could not be calculated for a single participant. | 4.5 (4.9) | 5.0 (13.0) | 5.0 (22.6) | 6.1 (11.7)
  SBP: PP Week 24 | 9.0 (1.4) | 10.0 (11.3) | 10.0 (4.2) | 14.0 (7.0) | 11.2 (5.9)
  DBP: GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
  DBP: GA Week 36 | -2.0 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 13.5 (2.1) | 3.0 (9.8) | 6.5 (23.3) | 5.9 (11.6)
  DBP: PP Week 24 | 6.5 (7.8) | 10.0 (2.8) | 8.0 (10.2) | 7.3 (11.8) | 7.8 (8.6)

28. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Weight at Baseline
Description: Absolute value of vital signs - body weight at baseline in maternal participants was reported.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Kilograms | 76.0 (29.7) | 64.0 (12.7) | 71.8 (8.8) | 75.8 (18.0) | 72.8 (16.7)

29. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Weight at GA Week 36
Description: Absolute value of vital signs -body weight at GA Week 36 in maternal participants was reported.
Time Frame: GA Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Kilograms | 130.6 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 77.6 (15.6) | 80.8 (7.9) | 87.3 (14.9) | 87.8 (19.9)

30. Primary Outcome: Maternal Participants: Absolute Value of Vital Signs - Body Weight at PP Week 24
Description: Absolute value of vital signs included body weight at PP Week 24 in maternal participants was reported.
Time Frame: PP Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Kilograms | 60.1 (8.0) | 69.5 (13.4) | 71.3 (11.1) | 78.0 (20.1) | 71.4 (14.3)

31. Primary Outcome: Maternal Participants: Change From Baseline in Vital Sign - Body Weight
Description: Change from baseline in vital signs- body weight in maternal participants was reported.
Time Frame: Baseline (GA Week 14), GA Week 36, and PP Week 24
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Kilograms
  GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
  GA Week 36 | 20.6 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 13.6 (3.0) | 8.6 (2.9) | 7.7 (1.4) | 11.1 (5.0)
  PP Week 24 | 1.0 (2.4) | 5.6 (0.8) | -0.5 (4.6) | 2.2 (2.9) | 1.7 (3.6)

32. Primary Outcome: Neonates/Infants: Absolute Value in Vital Signs - Body Temperature at Baseline
Description: Absolute value in vital signs parameter -body temperature at baseline was reported for all neonates/infants.
Time Frame: Baseline (PP Day 0)
Population: Neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'N' (overall number of participants analyzed) signifies number of neonates or infants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 3 | 2 | 10
Degree Celsius | 36.7 (0.4) | 36.8 (0.1) | 36.5 (0.1) | 36.7 (0.1) | 36.7 (0.2)

33. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Body Temperature at PP Week 1
Description: Absolute value of vital signs parameter -body temperature at PP Week 1 was reported for all neonates/infants.
Time Frame: PP Week 1
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 3 | 2 | 8
Degree Celsius | 37.1 (0.3) | 36.9 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 36.8 (0.1) | 37.1 (0.2) | 37.0 (0.2)

34. Primary Outcome: Neonates/Infants: Absolute Value in Vital Signs - Body Temperature at PP Week 4
Description: Absolute value in vital signs parameter - body temperature at PP Week 4 was reported for all neonates/infants.
Time Frame: PP Week 4
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 4 | 3 | 10
Degree Celsius | 36.8 (0.5) | 37.1 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 37.0 (0.5) | 37.2 (0.1) | 37.0 (0.4)

35. Primary Outcome: Neonates/Infants: Absolute Value in Vital Signs - Body Temperature at PP Week 24
Description: Absolute value in vital signs parameter -body temperature at PP Week 24 was reported for all neonates/infants.
Time Frame: PP Week 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 4 | 3 | 10
Degree Celsius | 36.5 (0.3) | 36.5 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 37.1 (0.4) | 37.5 (0.5) | 37.0 (0.5)

36. Primary Outcome: Neonates/Infants: Change From Baseline in Vital Signs - Body Temperature
Description: Change from baseline in vital signs- body temperature were reported for all neonates/infants.
Time Frame: Baseline (PP Day 0), PP Weeks 1, 4, and 24
Population: Neonates/infants analysis set: all live births to maternal participants who received at least 1 dose of nipocalimab. N (overall number of participants analyzed): number of neonate/infants evaluable, n (number analyzed): number of neonates/infants evaluable at specified timepoints. Only neonates/infants that had both baseline and post-baseline data available at a timepoint were analyzed. 2 participants with post-baseline but no baseline data were excluded.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 3 | 2 | 8
Degree Celsius
  PP Week 1: number analyzed (Participants) | 2 | 1 | 2 | 1 | 6
  PP Week 1 | 0.2 (0.4) | 0.1 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 0.3 (0.1) | 0.3 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 0.2 (0.2)
  PP Week 4 | 0.2 (0.1) | 0.4 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 0.6 (0.6) | 0.6 (0.1) | 0.5 (0.4)
  PP Week 24 | -0.4 (0.4) | -0.2 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 0.6 (0.5) | 1.0 (0.6) | 0.3 (0.7)

37. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Body Weight at Baseline
Description: Absolute value of vital signs parameter- body weight at baseline was reported for all neonates/infants.
Time Frame: Baseline (PP Day 0)
Population: Neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Kilograms | 2.4 (1.6) | 2.8 (0.4) | 2.8 (0.2) | 2.8 (0.4) | 2.7 (0.7)

38. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Body Weight at PP Week 1
Description: Absolute value of vital signs parameter - body weight at PP Week 1 was reported for all neonates/infants.
Time Frame: PP Week 1
Population: Neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'N' (overall number of participants analyzed) signifies the number of neonates or infants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 2 | 4 | 2 | 10
Kilograms | 1.6 (1.1) | 2.8 (0.5) | 2.7 (0.2) | 2.6 (0.3) | 2.5 (0.6)

39. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Body Weight at PP Week 4
Description: Absolute value of vital signs parameter - body weight at PP Week 4 was reported for all neonates/infants.
Time Frame: PP Week 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Kilograms | 2.6 (1.3) | 3.6 (1.1) | 3.4 (0.1) | 3.7 (0.7) | 3.3 (0.8)

40. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Body Weight at PP Week 24
Description: Absolute value of vital signs parameter - body weight at PP Week 24 was reported for all neonates/infants.
Time Frame: PP Week 24
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Kilograms | 6.4 (1.4) | 7.4 (1.6) | 7.6 (1.0) | 8.1 (0.6) | 7.4 (1.2)

41. Primary Outcome: Neonates/Infants: Change From Baseline in Vital Signs -Body Weight
Description: Change from baseline in vital signs - body weight were reported for all neonates/infants.
Time Frame: Baseline (PP Day 0), PP Weeks 1, 4, and 24
Population: Neonates/infants analysis set: all live births to maternal participants who received at least 1 dose of nipocalimab. 'n' (number analyzed): number of neonates/infants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Kilograms
  PP Week 1: number analyzed (Participants) | 2 | 2 | 4 | 2 | 10
  PP Week 1 | -0.1 (0.0) | 0.0 (0.1) | -0.1 (0.1) | -0.1 (0.1) | -0.1 (0.1)
  PP Week 4 | 0.2 (0.3) | 0.8 (0.7) | 0.6 (0.4) | 0.9 (0.3) | 0.6 (0.4)
  PP Week 24 | 4.0 (0.3) | 4.5 (1.2) | 4.8 (1.1) | 5.3 (0.8) | 4.7 (0.9)

42. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Respiratory Rate at Baseline
Description: Absolute value of vital signs parameter -respiratory rate at baseline was reported for all neonates/infants.
Time Frame: Baseline (PP Day 0)
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 2 | 4 | 2 | 10
Breaths per minute | 39.0 (7.1) | 47.0 (2.8) | 42.0 (5.2) | 49.5 (17.7) | 43.9 (8.1)

43. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Respiratory Rate at PP Week 1
Description: Absolute value of vital signs parameter - respiratory rate at PP Week 1 was reported for all neonates/infants.
Time Frame: PP Week 1
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 3 | 2 | 8
Breaths per minute | 36.0 (17.0) | 52.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 35.3 (1.2) | 54.0 (15.6) | 42.3 (12.7)

44. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Respiratory Rate at PP Week 4
Description: Absolute value of vital signs parameter - respiratory rate at PP Week 4 was reported for all neonates/infants.
Time Frame: PP Week 4
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 4 | 1 | 8
Breaths per minute | 69.0 (19.8) | 68.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 46.5 (5.5) | 40.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 54.0 (14.9)

45. Primary Outcome: Neonates/Infants: Absolute Value of Vital Signs - Respiratory Rate at PP Week 24
Description: Absolute value of vital signs parameter- respiratory rate at PP Week 24 was reported for all neonates/infants.
Time Frame: PP Week 24
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 4 | 3 | 10
Breaths per minute | 29.0 (9.9) | 32.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 45.3 (12.3) | 35.0 (7.8) | 37.6 (11.1)

46. Primary Outcome: Neonates/Infants: Change From Baseline in Vital Signs - Respiratory Rate
Description: Change from baseline in vital signs -respiratory rate was reported for all neonates/infants.
Time Frame: Baseline (PP Day 0), PP Weeks 1, 4, and 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 1 | 4 | 2 | 9
breaths per minute
  PP Week 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 6
  PP Week 1 | -10.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 3.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | -7.3 (7.0) | 6.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | -3.8 (8.0)
  PP Week 4: number analyzed (Participants) | 2 | 1 | 4 | 1 | 8
  PP Week 4 | 30.0 (26.9) | 23.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 4.5 (8.4) | 3.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 13.0 (16.9)
  PP Week 24: number analyzed (Participants) | 1 | 1 | 4 | 2 | 8
  PP Week 24 | -12.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | -13.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 3.3 (16.0) | -16.5 (27.6) | -5.6 (17.6)

47. Primary Outcome: Neonates/Infants: Absolute Value of Vital Sign - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Baseline
Description: Absolute value of vital signs parameter - SBP and DBP at baseline were reported for all neonates/infants.
Time Frame: Baseline (PP Day 0)
Population: Neonates/infants analysis set: all live births to maternal participants who received at least 1 dose of nipocalimab. Here, 'N' (overall number of participants analyzed): number of neonate/infants evaluable. N=0 in 'Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW' arm signifies that no data was collected because participants did not complete the scheduled assessments.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 0 | 2 | 2 | 7
Millimeters of mercury
  SBP | 73.7 (7.4) |  | 61.5 (19.1) | 61.5 (4.9) | 66.7 (11.2)
  DBP | 39.0 (2.6) |  | 32.0 (5.7) | 31.5 (7.8) | 34.9 (5.7)

48. Primary Outcome: Neonates/Infants: Absolute Value of Vital Sign - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at PP Week 1
Description: Absolute value of vital signs parameter - SBP and DBP at PP Week 1 were reported for all neonates/infants.
Time Frame: PP Week 1
Population: Neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'N' (overall number of participants analyzed) signifies the number of neonates or infants evaluable for this outcome measure. N=0 in 'Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW' arm signifies that no data was collected because participants did not complete the scheduled assessments.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 0 | 1 | 1 | 4
Millimeters of mercury
  SBP | 62.5 (2.1) |  | 75.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 65.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 66.3 (6.1)
  DBP | 50.0 (1.4) |  | 39.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 31.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant | 42.5 (9.3)

49. Primary Outcome: Neonates/Infants: Absolute Value of Vital Sign - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at PP Week 4
Description: Absolute value of vital signs parameter -SBP and DBP at PP Week 4 were reported for all neonates/infants.
Time Frame: PP Week 4
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 4
Millimeters of mercury
  SBP | 61.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 76.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 98.0 (4.2) | 83.3 (18.3)
  DBP | 31.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 30.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 59.0 (11.3) | 44.8 (17.7)

50. Primary Outcome: Neonates/Infants: Absolute Value of Vital Sign - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at PP Week 24
Description: Absolute value of vital signs parameter -SBP and DBP at PP Week 24 were reported for all neonates/infants.
Time Frame: PP Week 24
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 1 | 0 | 2 | 2 | 5
Millimeters of mercury
  SBP | 101.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 113.0 (36.8) | 103.5 (9.2) | 106.8 (19.8)
  DBP | 68.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 92.5 (26.2) | 58.0 (9.9) | 73.8 (22.4)

51. Primary Outcome: Neonates/Infants: Change From Baseline in Vital Signs - Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline in vital signs- SBP and DBP were reported for all neonates/infants.
Time Frame: Baseline (PP Day 0), PP Weeks 1, 4, and 24
Population: Neonates/infants analysis set was a use. N: number of neonate/infants evaluable, n (number analyzed): number of neonates/infants evaluable at specified timepoints. Only neonates/infants with both baseline and post-baseline data at a timepoint were analyzed. 2 participants with post-baseline but no baseline data were excluded. N=0 in 'Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW' arm signifies no data was collected because participants did not complete the scheduled assessments.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 2 | 0 | 1 | 2 | 5
Millimeters of mercury
  SBP: PP Week 1: number analyzed (Participants) | 2 | 0 | 1 | 1 | 4
  SBP: PP Week 1 | -7.0 (4.2) |  | 27.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 0.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 3.3 (16.4)
  SBP: PP Week 4: number analyzed (Participants) | 1 | 0 | 1 | 2 | 4
  SBP: PP Week 4 | -10.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 28.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 36.5 (9.2) | 22.8 (22.8)
  SBP: PP Week 24: number analyzed (Participants) | 1 | 0 | 1 | 1 | 3
  SBP: PP Week 24 | 33.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 39.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 52.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 41.3 (9.7)
  DBP: PP Week 1: number analyzed (Participants) | 2 | 0 | 1 | 1 | 4
  DBP: PP Week 1 | 11.5 (4.9) |  | 11.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | -6.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 7.0 (9.1)
  DBP: PP Week 4: number analyzed (Participants) | 1 | 0 | 1 | 2 | 4
  DBP: PP Week 4 | -10.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 2.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 27.5 (19.1) | 11.8 (21.8)
  DBP: PP Week 24: number analyzed (Participants) | 1 | 0 | 1 | 1 | 3
  DBP: PP Week 24 | 32.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. |  | 46.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 39.0 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 39.0 (7.0)

52. Primary Outcome: Percentage of Maternal Participants With Intrauterine Growth Restriction (IUGR) Based on Ultrasound Assessments
Description: Percentage of maternal participants with intrauterine growth restriction (IUGR) based on ultrasound assessments and guidelines from American College of Obstetricians and Gynecologists, and Society for Maternal-Fetal Medicine was reported. This outcome measure provided the incidence of with IUGR at delivery. IUGR is defined as weight below the 10th percentile for gestational age based on the World Health Organization (WHO) fetal growth curve.
Time Frame: Baseline (GA Week 14), GA Weeks 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, and 36
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, n (number analyzed) signifies number of participants evaluable at specified timepoints and n=0 signifies that no participants were available for the analysis.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Percentage of maternal participants
  Baseline: number analyzed (Participants) | 2 | 0 | 3 | 3 | 8
  Baseline | 0 |  | 0 | 0 | 0
  GA Week 16: number analyzed (Participants) | 1 | 2 | 3 | 4 | 10
  GA Week 16 | 0 | 0 | 0 | 0 | 0
  GA Week 18: number analyzed (Participants) | 1 | 2 | 4 | 4 | 11
  GA Week 18 | 0 | 0 | 0 | 0 | 0
  GA Week 20: number analyzed (Participants) | 2 | 1 | 4 | 4 | 11
  GA Week 20 | 50.0 | 0 | 0 | 0 | 9.1
  GA Week 22: number analyzed (Participants) | 2 | 1 | 4 | 3 | 10
  GA Week 22 | 0 | 0 | 0 | 0 | 0
  GA Week 24: number analyzed (Participants) | 3 | 1 | 4 | 3 | 11
  GA Week 24 | 0 | 0 | 0 | 0 | 0
  GA Week 26: number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
  GA Week 26 | 0 | 50.0 | 0 | 0 | 8.3
  GA Week 28: number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
  GA Week 28 | 0 | 50.0 | 0 | 0 | 8.3
  GA Week 30: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  GA Week 30 | 0 | 0 | 0 | 0 | 0
  GA Week 32: number analyzed (Participants) | 2 | 1 | 4 | 3 | 10
  GA Week 32 | 0 | 100.0 | 0 | 0 | 10.0
  GA Week 34: number analyzed (Participants) | 2 | 1 | 4 | 2 | 9
  GA Week 34 | 0 | 0 | 0 | 0 | 0
  GA Week 36: number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
  GA Week 36 | 0 | 0 | 0 | 0 | 0

53. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: Amniotic Fluid Index (AFI) at Baseline
Description: Percentage of maternal participants with abnormal amniotic fluid values: amniotic fluid index (AFI) at baseline was reported. The amniotic fluid volume abnormality was categorized as an AFI <5 centimeter (cm) or >24 cm.
Time Frame: Baseline (GA Week 14)
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies the number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Percentage of maternal participants | 0 | 50.0 | 50.0 | 0 | 25.0

54. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: AFI at GA Week 26
Description: Percentage of maternal participants with abnormal amniotic fluid values: AFI at GA Week 26 was reported. The amniotic fluid volume abnormality was categorized as an AFI <5 cm or >24 cm.
Time Frame: GA Week 26
Population: The FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies the number of participants evaluable for this outcome measure. Data was not collected and analyzed for Group 2 as no participant was available for the analysis at the specified timepoint.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 0 | 4 | 3 | 8
Percentage of maternal participants | 0 |  | 25.0 | 0 | 12.5

55. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: AFI at GA Week 36
Description: Percentage of maternal participants with abnormal amniotic fluid values: AFI at GA Week 36 was reported. The amniotic fluid volume abnormality was categorized as an AFI <5 cm or >24 cm.
Time Frame: GA Week 36
Population: as for outcome 53
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 1 | 3 | 2 | 7
Percentage of maternal participants | 0 | 0 | 33.3 | 0 | 14.3

56. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: Maximum Vertical Pocket (MVP) at Baseline
Description: Percentage of maternal participants with abnormal amniotic fluid values: maximum vertical pocket (MVP) at baseline was reported. The amniotic fluid volume abnormality was categorized as MVP <2 cm or >8 cm.
Time Frame: From Baseline (GA Week 14)
Population: as for outcome 53
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 9
Percentage of maternal participants | 0 | 0 | 0 | 0 | 0

57. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: MVP at GA Week 18
Description: Percentage of maternal participants with abnormal amniotic fluid values: MVP at GA Week 18 was reported. The amniotic fluid volume abnormality was categorized as MVP <2 cm or >8 cm.
Time Frame: GA Week 18
Population: as for outcome 53
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
Percentage of maternal participants | 0 | 0 | 0 | 25.0 | 8.3

58. Primary Outcome: Percentage of Maternal Participants With Abnormal Amniotic Fluid Values: MVP at GA Week 22
Description: Percentage of maternal participants with abnormal amniotic fluid values: MVP at GA Week 22 was reported. The amniotic fluid volume abnormality was categorized as MVP <2 cm or >8 cm.
Time Frame: GA Week 22
Population: as for outcome 53
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Percentage of maternal participants | 0 | 0 | 0 | 0 | 0

59. Primary Outcome: Number of Neonates/Infants With Appearance, Pulse, Grimace Response, Activity, Respiration (Apgar) Score
Description: Number of neonates/infants with Apgar score from 1 to 10 minutes of life were reported. The system provided a standardized assessment for infants after delivery. The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2. The score is reported at 1 minute and 5 minutes after birth for all infants, and at 5-minute intervals thereafter until 20 minutes for infants with a score less than 7. This is using an Apgar scale which ranges from minimum total score of 0 and maximum total score of 10, with higher score representing a better outcome.
Time Frame: 1, 5, and 10 minutes after birth at PP Day 0
Population: Neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, n (number analyzed): number of neonates or infants evaluable for each arm at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants
  1 minute: <5 Score | 1 | 0 | 0 | 1 | 2
  1 minute: 5-7 Score | 0 | 0 | 1 | 0 | 1
  1 minute: 8-10 Score | 2 | 2 | 3 | 2 | 9
  5 minute: <5 Score | 0 | 0 | 0 | 0 | 0
  5 minute: 5-7 Score | 0 | 0 | 0 | 1 | 1
  5 minute: 8-10 Score | 3 | 2 | 4 | 2 | 11
  10 minute: <5 Score: number analyzed (Participants) | 1 | 2 | 2 | 2 | 7
  10 minute: <5 Score | 0 | 0 | 0 | 0 | 0
  10 minute: 5-7 Score: number analyzed (Participants) | 1 | 2 | 2 | 2 | 7
  10 minute: 5-7 Score | 0 | 0 | 0 | 1 | 1
  10 minute: 8-10 Score: number analyzed (Participants) | 1 | 2 | 2 | 2 | 7
  10 minute: 8-10 Score | 1 | 2 | 2 | 1 | 6

60. Primary Outcome: Number of Maternal Participants With Concomitant Medications and Therapies
Description: Number of maternal participants with concomitant medications and therapies were reported.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to PP Week 24 (up to 50 weeks)
Population: Safety analysis set included all maternal participants who received at least 1 dose of nipocalimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Participants | 3 | 2 | 4 | 4 | 13

61. Primary Outcome: Number of Neonates/Infants With Concomitant Medications and Therapies
Description: Number of neonates/infants with concomitant medications and therapies were reported.
Time Frame: From birth (PP Day 0) up to PP Week 96
Population: The neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Participants | 3 | 2 | 4 | 3 | 12

62. Primary Outcome: Percentage of Maternal Participants With Live Birth at or After Gestational Age (GA) Week 32 and Without an Intrauterine Transfusion (IUT) Throughout Their Entire Pregnancies
Description: Percentage of maternal participants with live birth at or after GA Week 32 and without an IUT throughout their entire pregnancies were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Number (95% Confidence Interval); unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kgTAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Percentage of maternal participants | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 75.0 [19.4 to 99.4] | 50.0 [6.8 to 93.2] | 53.8 [25.1 to 80.8]

63. Secondary Outcome: Percentage of Maternal Participants With Live Birth
Description: Percentage of maternal participants with live birth were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Percentage of maternal participants | 100 | 100 | 100 | 75 | 92.3

64. Secondary Outcome: Percentage of Maternal Participants Without an Intrauterine Transfusion (IUT) Before Gestational Age (GA) Week 24
Description: Percentage of maternal participants without an IUT before GA Week 24 were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 24
Population: FAS included all maternal participants who received any dose of nipocalimab.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Percentage of maternal participants | 100 | 100 | 100 | 75 | 92.3

65. Secondary Outcome: Maternal Participants : Gestational Age (GA) at First Intrauterine Transfusion (IUT)
Description: Gestational age (GA) at first IUT for maternal participants were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: as for outcome 8
Measure: Median (Full Range); unit: weeks
Groups:
- Group 1 (Maternal): 30 mg/kg BLW: Maternal subjects received a single dose intravenous (IV) infusion of nipocalimab 30 milligrams per kilograms (mg/kg) based on baseline weight (BLW), once weekly from gestation age (GA) Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal subjects were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [Postpartum {PP} Week 24]).
- Group 2 (Maternal): 30 to 45 mg/kg BLW: Maternal subjects received a single dose of IV infusion of nipocalimab 30 mg/kg initially based on BLW followed by nipocalimab 45 mg/kg with increase in weight, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal subjects were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 3 (Maternal): 45 mg/kg BLW: Maternal subjects received a single dose IV infusion of nipocalimab 45 mg/kg based on BLW, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal subjects were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 4 (Maternal): 45 mg/kg TAW: Maternal subjects received a single dose IV infusion of nipocalimab 45 mg/kg based on time-adjusted weight (TAW), once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal subjects were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- All Maternal Subjects: Maternal subjects of Group 1 (30 milligrams per kilograms [mg/kg] baseline weight [BLW]), Group 2 (30 to 45 mg/kg BLW), Group 3 (45 mg/kg BLW), and Group 4 (45 mg/kg time-adjusted weight [TAW]) who received a single dose of intravenous (IV) infusions of nipocalimab once weekly from gestation age (GA) Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal subjects were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Subjects
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 6
weeks | 25 [24 to 25] | 28 [28 to 28] | 29 [29 to 29] | 27 [22 to 31] | 27 [22 to 31]

66. Secondary Outcome: Median Number of Intrauterine Transfusion (IUT) Per Maternal Participant
Description: Median number of intrauterine transfusion (IUT) per maternal participants were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Median (Full Range); unit: IUTs per maternal participant
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
IUTs per maternal participant | 4 [3 to 5] | 5 [5 to 5] | 3 [3 to 3] | 1 [1 to 1] | 3 [1 to 5]

67. Secondary Outcome: Frequency of Intrauterine Transfusions (IUTs) on Maternal Participants
Description: Frequency of intrauterine transfusions (IUTs) on maternal participants were reported. Frequency of IUTs was defined as total number of IUTs divided by the (date of delivery - date of first IUT +1)/7.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: The FAS included all maternal participants who received any dose of nipocalimab.
Measure: Median (Full Range); unit: IUT/week
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
IUT/week | 0.52 [0.48 to 0.57] | 0.56 [0.56 to 0.56] | 0.43 [0.43 to 0.43] | 0.70 [0.64 to 0.78] | 0.56 [0.43 to 0.78]

68. Secondary Outcome: Percentage of Maternal Participants With Fetal Hydrops in Utero or Post Birth
Description: Percentage of maternal participants with fetal hydrops in utero or post birth were reported.
Time Frame: From baseline (Gestational Age [GA] Week 14) up to PP Week 24 (up to 50 weeks)
Population: FAS included all maternal participants who received any dose of nipocalimab. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of maternal participants
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Percentage of maternal participants | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 26.5]

69. Secondary Outcome: Maternal Participants: Gestational Age at Time of Delivery
Description: Gestational age at time of delivery for maternal participants were reported.
Time Frame: From baseline (GA Week 14) up to GA Week 37
Population: FAS included all maternal participants who received any dose of nipocalimab.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
Weeks | 36 [29 to 37] | 36 [35 to 37] | 36 [36 to 37] | 35 [23 to 37] | 36 [23 to 37]

70. Secondary Outcome: Percentage of Neonates Who Required Phototherapy
Description: Percentage of neonates who required phototherapy were reported.
Time Frame: From birth (PP Day 0) up to PP Week 24
Population: as for outcome 61
Measure: Number; unit: Percentage of neonates
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Percentage of neonates | 100 | 50 | 100 | 100 | 91.7

71. Secondary Outcome: Percentage of Neonates Who Required Exchange Transfusions
Description: Percentage of neonates who required exchange transfusions were reported.
Time Frame: From birth (PP Day 0) up to PP Week 24
Population: as for outcome 61
Measure: Number; unit: Percentage of neonates
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Percentage of neonates | 0 | 0 | 0 | 33.3 | 8.3

72. Secondary Outcome: Duration of Postnatal Phototherapy Required by Neonates
Description: Duration of postnatal phototherapy required by neonates were reported.
Time Frame: From birth (PP Day 0) up to PP Week 24
Population: The neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 1 | 4 | 3 | 11
hours | 96.0 [84.00 to 301.07] | 46.68 [46.68 to 46.68] | 100.87 [12.00 to 173.95] | 86.98 [72.00 to 127.33] | 86.98 [12.00 to 301.07]

73. Secondary Outcome: Percentage of Neonates Who Required Simple Transfusions in the First 12 Weeks of Life
Description: Percentage of neonates who required simple transfusions in the first 12 weeks of life were reported.
Time Frame: From birth (PP Day 0) up to PP Week 12
Population: as for outcome 61
Measure: Number; unit: Percentage of neonates
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Percentage of neonates | 66.7 | 50.0 | 50.0 | 33.3 | 50.0

74. Secondary Outcome: Number of Simple Transfusions Required by Neonate in the First 12 Weeks of Life
Description: Number of simple transfusions required by neonate in the first 12 weeks of life were reported.
Time Frame: From birth (PP Day 0) up to PP Week 12
Population: as for outcome 61
Measure: Median (Full Range); unit: Simple transfusions
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Simple transfusions | 4.5 [3. to 6] | 4.0 [4 to 4] | 1.0 [1 to 1] | 1.0 [1 to 1] | 2.0 [1 to 6]

75. Secondary Outcome: Maternal Serum Unoccupied Neonatal Concentration of Participants Fc Receptor [FcRn] Receptor Occupancy (RO) in Monocytes by Nipocalimab
Description: Maternal serum unoccupied neonatal concentration of Participants Fc Receptor [FcRn] receptor occupancy (RO) in Monocytes by nipocalimab were reported.
Time Frame: Baseline (GA Week 14), GA Week 16, GA Week 36, PP Day 0, PP Week 4, and PP Week 24
Population: The pharmacodynamics (PD) evaluable analysis set included all maternal participants who received at least 1 dose of nipocalimab and had at least 1 valid post-dose PD (RO or IgG) assessment. Here, ''n' (number analyzed) signifies number of participants evaluable for specified timepoints. Here, n = 0 indicates that no laboratory measurements were collected at that specific time point as no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: percentage of receptors unoccupied
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
percentage of receptors unoccupied
  Baseline | 100.00 (0.000) | 100.00 (0.000) | 100.00 (0.000) | 100.00 (0.000) | 100.00 (0.000)
  GA Week 16: number analyzed (Participants) | 3 | 2 | 3 | 4 | 12
  GA Week 16 | 2.80 (0.346) | 2.50 (1.556) | 4.20 (3.816) | -0.15 (6.276) | 2.12 (4.103)
  GA Week 36: number analyzed (Participants) | 1 | 1 | 2 | 2 | 6
  GA Week 36 | 12.20 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 3.80 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 5.40 (1.838) | 3.75 (1.202) | 5.72 (3.420)
  PP Day 0: number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
  PP Day 0 | 126.75 (6.859) | 21.00 (22.486) | 68.83 (43.253) | 39.30 (43.856) | 60.67 (48.532)
  PP Week 4: number analyzed (Participants) | 2 | 0 | 4 | 4 | 10
  PP Week 4 | 107.55 (68.943) |  | 130.78 (49.901) | 121.55 (54.002) | 122.44 (49.09)
  PP Week 24: number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
  PP Week 24 | 99.60 (5.091) | 98.45 (15.486) | 114.15 (28.333) | 117.20 (29.816) | 110.13 (23.549)

76. Secondary Outcome: Serum Unoccupied Concentration of Participants Fc Receptor [FcRn] Receptor Occupancy (RO) in Monocytes of Neonate by Nipocalimab
Description: Serum unoccupied FcRn RO in monocytes of neonate by Nipocalimab were reported.
Time Frame: From birth (PP Day 0) up to PP Week 24
Population: The PD evaluable set neonates included all neonate/infant participants who had at least 1 valid PD (RO or IgG) assessment. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of receptors unoccupied
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
percentage of receptors unoccupied | 118.20 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 70.60 (19.233) | 80.87 (18.029) | 74.50 (33.093) | 81.38 (23.295)

77. Secondary Outcome: Maternal Participants: Change From Baseline in Serum Concentration of Total Immunoglobulin G (IgG) and Subclasses (IgG1, IgG2, IgG3, IgG4), IgA, IgM, and IgE
Description: Change from baseline in serum concentration of total immunoglobulin G (IgG) and subclasses (IgG1, IgG2, IgG3, IgG4), IgA, IgM, and IgE were reported.
Time Frame: IgG: Baseline (GA Week 14), GA Week 16, GA Week 36, birth (PP Day 0), PP Week 4, and PP Week 24; IgG1, IgG2, IgG3, IgG4, IgA, IgM, and IgE: baseline (GA Week 14), GA Week 36
Population: Pharmacodynamics (PD) evaluable analysis set included all maternal participants who received at least 1 dose of nipocalimab and had at least 1 valid post-dose PD (RO or IgG) assessment. Here, 'n' (number analyzed) signifies number of participants evaluable at each timepoint for respective category. Here, n = 0 indicates that no laboratory measurements were collected at that specific time point as no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: grams/liter (g/L)
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW | All Maternal Participants
Number analyzed (Participants) | 3 | 2 | 4 | 4 | 13
grams/liter (g/L)
  IgG: GA Week 16 | -8.12 (2.235) | -7.31 (0.813) | -6.51 (1.285) | -8.19 (1.018) | -7.52 (1.464)
  IgG: GA Week 36: number analyzed (Participants) | 2 | 2 | 4 | 3 | 11
  IgG: GA Week 36 | -7.52 (1.549) | -5.26 (2.574) | -5.83 (2.380) | -8.34 (1.305) | -6.72 (2.146)
  IgG: birth (PP Day 0): number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
  IgG: birth (PP Day 0) | -0.40 (0.884) | -2.64 (0.148) | -2.45 (1.016) | -4.38 (2.771) | -2.78 (2.111)
  IgG: PP Week 4: number analyzed (Participants) | 2 | 0 | 4 | 4 | 10
  IgG: PP Week 4 | 1.88 (1.803) |  | -0.17 (0.638) | 1.10 (3.455) | 0.75 (2.277)
  IgG: PP Week 24: number analyzed (Participants) | 2 | 2 | 4 | 4 | 12
  IgG: PP Week 24 | 2.56 (0.255) | 2.02 (0.622) | 1.34 (0.411) | 2.61 (1.101) | 2.08 (0.873)
  IgG1: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgG1: GA Week 36 | -4.35 (1.386) | -3.94 (1.464) | -3.45 (1.421) | -5.46 (1.006) | -4.33 (1.356)
  IgG2: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgG2: GA Week 36 | -2.48 (0.085) | -1.29 (0.629) | -1.91 (1.013) | -2.31 (1.192) | -2.02 (0.888)
  IgG3: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgG3: GA Week 36 | -0.25 (0.045) | -0.23 (0.228) | -0.24 (0.195) | -0.38 (0.124) | -0.28 (0.151)
  IgG4: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgG4: GA Week 36 | -0.39 (0.209) | -0.06 (0.045) | -0.13 (0.066) | -0.28 (0.140) | -0.21 (0.163)
  IgA: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgA: GA Week 36 | 0.17 (0.163) | 0.11 (0.191) | 0.20 (0.382) | 0.05 (0.015) | 0.13 (0.208)
  IgM: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgM: GA Week 36 | 0.01 (0.120) | -0.06 (0.049) | 0.01 (0.072) | -0.12 (0.075) | -0.04 (0.087)
  IgE: GA Week 36: number analyzed (Participants) | 2 | 2 | 3 | 3 | 10
  IgE: GA Week 36 | -0.31 (0.420) | 0.00 (0.003) | 0.01 (0.012) | 0.00 (0.086) | -0.06 (0.197)

78. Secondary Outcome: Neonates/Infants: Change From Baseline in Serum Concentration of Total IgG, IgA, IgM, and IgE
Description: Change from baseline in serum concentration of total IgG, IgA, IgM, and IgE were reported in neonates/infants were reported.
Time Frame: Baseline (PP Day 0), PP Weeks 4, 24, 96
Population: PD evaluable set - neonates included all neonate/infant participants who had at least 1 valid PD (RO or IgG) assessment. Here, 'n' (number analyzed): number of neonates or infants evaluable for each arm at specified time points. Here, n = 0 indicates that no laboratory measurements were collected at that specific time point as no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: grams/liter (g/L)
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
grams/liter (g/L)
  IgG: PP Week 4: number analyzed (Participants) | 1 | 1 | 3 | 2 | 7
  IgG: PP Week 4 | 4.61 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -2.16 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.37 (2.521) | -0.87 (0.559) | 0.26 (2.594)
  IgG: PP Week 24: number analyzed (Participants) | 1 | 1 | 4 | 1 | 7
  IgG: PP Week 24 | -7.59 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -0.09 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.78 (2.675) | 1.68 (NA) — "NA" signifies that SD could not be calculated for a single participant. | -0.41 (3.723)
  IgG: PP Week 96: number analyzed (Participants) | 0 | 1 | 3 | 2 | 6
  IgG: PP Week 96 |  | -1.41 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 5.55 (2.866) | 4.62 (1.683) | 4.08 (3.361)
  IgA: PP Week 4: number analyzed (Participants) | 1 | 0 | 2 | 1 | 4
  IgA: PP Week 4 | 0.00 (NA) — "NA" signifies that SD could not be calculated for a single participant. |  | 0.00 (0.000) | 0.03 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.01 (0.015)
  IgA: PP Week 24: number analyzed (Participants) | 1 | 1 | 3 | 1 | 6
  IgA: PP Week 24 | 0.02 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.07 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.23 (0.127) | -0.87 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.15 (0.121)
  IgA: PP Week 96: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5
  IgA: PP Week 96 |  | 0.28 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.47 (0.297) | 0.29 (0.035) | 0.36 (0.181)
  IgM: PP Week 4: number analyzed (Participants) | 1 | 0 | 2 | 2 | 5
  IgM: PP Week 4 | 0.10 (NA) — "NA" signifies that SD could not be calculated for a single participant. |  | 0.17 (0.092) | 0.34 (0.071) | 0.22 (0.125)
  IgM: PP Week 24: number analyzed (Participants) | 1 | 1 | 3 | 1 | 6
  IgM: PP Week 24 | 0.32 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.26 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.61 (0.078) | 0.44 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.48 (0.166)
  IgM: PP Week 96: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5
  IgM: PP Week 96 |  | 0.53 (NA) — "NA" signifies that SD could not be calculated for a single participant.. | 1.04 (0.014) | 0.86 (0.368) | 0.87 (0.278)
  IgE: PP Week 4: number analyzed (Participants) | 1 | 0 | 3 | 2 | 6
  IgE: PP Week 4 | 0.00 (NA) — "NA" signifies that SD could not be calculated for a single participant. |  | 0.00 (0.007) | 0.00 (0.000) | 0.00 (0.004)
  IgE: PP Week 24: number analyzed (Participants) | 1 | 1 | 3 | 1 | 6
  IgE: PP Week 24 | 0.01 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.00 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.03 (0.059) | 0.02 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.02 (0.040)
  IgE: PP Week 96: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5
  IgE: PP Week 96 |  | 0.02 (NA) — "NA" signifies that SD could not be calculated for a single participant. | 0.02 (0.008) | 0.03 (0.027) | 0.02 (0.016)

79. Secondary Outcome: Serum Concentrations of Nipocalimab in Maternal Participants
Description: Serum concentrations of Nipocalimab in maternal participants were reported.
Time Frame: Pre dose and post dose: GA Week 14 and GA Week 24; Birth (PP Day 0), PP Week 4 and PP Week 24
Population: Pharmacokinetic evaluable analysis set included all maternal participants who received at least 1 dose of nipocalimab and had at least 1 valid post-dose blood sample drawn for PK analysis. Here, 'n' (number analyzed) signifies number of participants evaluable for specified timepoints. Here, n = 0 indicates that no laboratory measurements were collected at that specific time point as no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Group 1 (Maternal): 30 mg/kg BLW | Group 2 (Maternal): 30 to 45 mg/kg BLW | Group 3 (Maternal): 45 mg/kg BLW | Group 4 (Maternal): 45 mg/kg TAW
Number analyzed (Participants) | 3 | 2 | 4 | 4
mcg/mL
  GA Week 14: Pre-dose | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  GA Week 14: Post-dose | 726.00 (138.01) | 577.00 (110.31) | 947.75 (193.17) | 928.50 (159.05)
  GA Week 24: Pre-dose: number analyzed (Participants) | 2 | 2 | 4 | 3
  GA Week 24: Pre-dose | 58.25 (43.63) | 71.15 (19.87) | 197.25 (73.27) | 205.00 (82.18)
  GA Week 24: Post-dose: number analyzed (Participants) | 2 | 2 | 4 | 3
  GA Week 24: Post-dose | 736.50 (101.12) | 629.00 (90.51) | 1051.25 (196.49) | 1246.67 (202.32)
  PP Day 0: number analyzed (Participants) | 2 | 1 | 3 | 4
  PP Day 0 | 0.01 (0.02) | 100.0 (NA) — SD could not be calculated for a single participant. | 14.54 (25.16) | 278.96 (547.41)
  PP Week 4: number analyzed (Participants) | 2 | 0 | 4 | 4
  PP Week 4 | 0.00 (0.00) |  | 0.00 (0.00) | 0.00 (0.00)
  PP Week 24: number analyzed (Participants) | 2 | 2 | 4 | 3
  PP Week 24 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

80. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Total and Sub Scale Score in Neonates/Infants
Description: The 45-item PedsQL infant Scales (ages 13-24 months) included physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning. Health summary score for psychosocial (sum of all items over number of items: emotional, social, cognitive functioning scales) and physical (sum of the items over number of items: physical functioning and symptoms scales), as well as a total score (sum of all items over number of items answered on all scales). Items were reverse-scored and linearly transformed to 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0). PedsQL a validated scale ranging from 0 -100, higher scores = a better quality of life.
Time Frame: PP Week 96
Population: The neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'N' overall (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 8
Score on a scale
  Overall Total Score | 86.67 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 86.67 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 88.15 (13.95) | 84.44 (6.26) | 86.39 (8.35)
  Psychosocial Health Total Score | 78.85 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 88.46 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 86.86 (15.21) | 77.88 (8.22) | 82.69 (10.47)
  Physical Health Total Score | 97.37 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 84.21 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 89.91 (12.23) | 93.42 (8.22) | 91.45 (8.78)
  Physical Functioning Score | 100.00 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 88.89 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 90.74 (16.04) | 96.30 (3.21) | 93.75 (9.59)
  Physical Symptoms Score | 95.00 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 80.00 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 89.17 (10.10) | 90.83 (13.77) | 89.38 (10.07)
  Emotional Functioning Score | 62.50 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 95.83 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 81.25 (17.80) | 70.83 (7.22) | 76.82 (14.50)
  Social Functioning Score | 100.00 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 100.00 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 91.67 (14.43) | 95.00 (8.66) | 95.00 (9.64)
  Cognitive Functioning Score | 88.89 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 72.22 (NA) — "NA" signifies that standard deviation (SD) could not be calculated for a single participant. | 91.67 (14.43) | 77.78 (12.11) | 83.68 (12.90)

81. Secondary Outcome: Ages and Stages Questionnaires, Third Edition (ASQ-3) Total Domain Score in Neonates/Infants
Description: The ASQ-3 assesses young child's (2-66 months) development based on age and included 6 questions in each area of child development: communication, gross motor, fine motor, problem solving, and personal-social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3 and each domain score could range from 0 to 60 points which higher score signifying stronger development.
Time Frame: At PP 6 month, PP 12 month, and PP 24 month
Population: The neonates/infants analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. Here, 'n': number of participants evaluable for each arm at specific time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW | All Neonates and Infants
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 12
Score on a scale
  Communication Total Score: PP 6-month | 36.7 (5.8) | 40.0 (7.1) | 48.8 (6.3) | 51.7 (2.9) | 45.0 (8.0)
  Communication Total Score: PP 12-month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Communication Total Score: PP 12-month | 45.0 (15.0) | 40.0 (7.1) | 43.3 (11.5) | 40.0 (10.0) | 42.3 (10.1)
  Communication Total Score: PP 24-month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Communication Total Score: PP 24-month | 45.0 (15.0) | 37.5 (24.7) | 48.3 (2.9) | 26.7 (2.9) | 39.5 (13.9)
  Gross Motor Total Score: PP 6-month | 35.0 (10.0) | 22.5 (3.5) | 30.0 (9.1) | 25.0 (13.2) | 28.8 (9.8)
  Gross Motor Total Score: PP 12-month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Gross Motor Total Score: PP 12-month | 31.7 (17.6) | 40.0 (28.3) | 21.7 (18.9) | 23.3 (23.6) | 28.2 (19.4)
  Gross Motor Total Score: PP 24-month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Gross Motor Total Score: PP 24-month | 43.3 (17.6) | 60.0 (0.0) | 50.0 (8.7) | 56.7 (2.9) | 51.8 (11.0)
  Fine Motor Total Score: PP 6-Month | 26.7 (7.6) | 35.0 (21.2) | 43.8 (8.5) | 35.0 (18.0) | 35.8 (13.3)
  Fine Motor Total Score: PP 12-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Fine Motor Total Score: PP 12-Month | 46.7 (2.9) | 57.5 (3.5) | 50.0 (0.0) | 36.7 (7.6) | 46.8 (8.4)
  Fine Motor Total Score: PP 24-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Fine Motor Total Score: PP 24-Month | 50.0 (10.0) | 47.5 (3.5) | 55.0 (8.7) | 50.0 (5.0) | 50.9 (7.0)
  Problem Solving Total Score: PP 6-Month | 40.0 (10.0) | 37.5 (17.7) | 38.8 (11.1) | 26.7 (10.4) | 35.8 (11.4)
  Problem Solving Total Score: PP 12-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Problem Solving Total Score: PP 12-Month | 23.3 (15.3) | 25.0 (7.1) | 41.7 (2.9) | 40.0 (8.7) | 33.2 (12.1)
  Problem Solving Total Score: PP 24-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Problem Solving Total Score: PP 24-Month | 48.3 (7.6) | 37.5 (17.7) | 35.0 (8.7) | 41.7 (2.9) | 40.9 (9.4)
  Personal-Social Total Score: PP 6-Month | 43.3 (5.8) | 30.0 (7.1) | 40.0 (10.8) | 20.0 (13.2) | 34.2 (12.9)
  Personal-Social Total Score: PP 12-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Personal-Social Total Score: PP 12-Month | 21.7 (2.9) | 37.5 (3.5) | 35.0 (5.0) | 30.0 (20.0) | 30.5 (11.3)
  Personal-Social Total Score: PP24-Month: number analyzed (Participants) | 3 | 2 | 3 | 3 | 11
  Personal-Social Total Score: PP24-Month | 48.3 (10.4) | 45.0 (21.2) | 50.0 (13.2) | 50.0 (5.0) | 48.6 (10.5)

ADVERSE EVENTS:
Time Frame: All-cause mortality: Maternal: Screening (GA Week 8) up to PP Week 24 (up to 56 weeks), Neonates/Infants: Birth (PP Day 0) up to PP Week 96; SAE and other AEs: Maternal: From baseline (GA Week 14) up to PP Week 24 (up to 50 weeks), Neonates/Infants: From birth (PP Day 0) up to PP Week 96
Description: Maternal: Safety analysis set included all maternal participants who have received at least 1 dose of nipocalimab. Neonates/Infants: Safety analysis set included all live births to maternal participants who received at least 1 dose of nipocalimab in the study pregnancy. For Group 2, pooled data for 30 mg/kg and 45 mg/kg was collected and analyzed as exposure to 30 mg/kg was very limited with minimal cumulative dosing and sample size was too small for meaningful separate analysis.
Groups:
- Group 1 (Maternal): 30mg/kg BLW: Maternal participants received a single dose intravenous (IV) infusion of nipocalimab 30 milligrams per kilograms (mg/kg) based on baseline weight (BLW), once weekly from gestation age (GA) Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [Postpartum {PP} Week 24]).
- Group 2 (Maternal): 30 to45 mg/kg BLW: Maternal participants received a single dose IV infusion of nipocalimab 30 mg/kg initially based on BLW followed by nipocalimab 45 mg/kg with increase in weight, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 3 (Maternal): 45mg/kg BLW: Maternal participants received a single dose IV infusion of nipocalimab 45 mg/kg based on BLW, once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
- Group 4 (Maternal): 45mg/kg TAW: Maternal participants received a single dose IV infusion of nipocalimab 45 mg/kg based on time-adjusted weight (TAW), once weekly from GA Week 14 to GA Week 35. The first infusion of nipocalimab was administered over 60 minutes, subsequent infusions were administered over 30 minutes. Maternal participants were followed up for safety during the safety follow up period of 24 weeks after delivery at approximately GA Week 37 (up to Week 61 [PP Week 24]).
Arm/Group | Group 1 (Maternal): 30mg/kg BLW | Group 2 (Maternal): 30 to45 mg/kg BLW | Group 3 (Maternal): 45mg/kg BLW | Group 4 (Maternal): 45mg/kg TAW | Group 1 (Neonates and Infants): 30 mg/kg BLW | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW | Group 3 (Neonates and Infants): 45 mg/kg BLW | Group 4 (Neonates and Infants): 45 mg/kg TAW
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/4 | 0/4 | 0/3 | 0/2 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/2 | 1/4 | 2/4 | 2/3 | 1/2 | 1/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 4/4 | 4/4 | 3/3 | 2/2 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Maternal): 30mg/kg BLW (N=3) | Group 2 (Maternal): 30 to45 mg/kg BLW (N=2) | Group 3 (Maternal): 45mg/kg BLW (N=4) | Group 4 (Maternal): 45mg/kg TAW (N=4) | Group 1 (Neonates and Infants): 30 mg/kg BLW (N=3) | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW (N=2) | Group 3 (Neonates and Infants): 45 mg/kg BLW (N=4) | Group 4 (Neonates and Infants): 45 mg/kg TAW (N=3)
Anaemia Neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Foetal Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foetal Heart Rate Deceleration Abnormality (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia Neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foetal Growth Restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature Separation of Placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retained Placenta or Membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subchorionic Haematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Maternal): 30mg/kg BLW (N=3) | Group 2 (Maternal): 30 to45 mg/kg BLW (N=2) | Group 3 (Maternal): 45mg/kg BLW (N=4) | Group 4 (Maternal): 45mg/kg TAW (N=4) | Group 1 (Neonates and Infants): 30 mg/kg BLW (N=3) | Group 2 (Neonates and Infants): 30 to 45 mg/kg BLW (N=2) | Group 3 (Neonates and Infants): 45 mg/kg BLW (N=4) | Group 4 (Neonates and Infants): 45 mg/kg TAW (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Anaemia Neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Foetal Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinopathy of Prematurity (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion Site Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Puncture Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Biliary Colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-Alcoholic Fatty Liver (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asymptomatic Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial Vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1
Otitis Media Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Immunoglobulin G Decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Blood Potassium Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein Total Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reticulocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid Intake Reduced (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foetal Hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Premature Separation of Placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small for Dates Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine Contractions During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Social Anxiety Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pruritus Allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Scar Pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Caesarean Section (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epidural Anaesthesia (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Superficial Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Substantial contributions to the conception or design of the work; or the acquisition, analysis, or interpretation of data for the work; AND Drafting the work or revising it critically for important intellectual content; AND Final approval of the version to be published; AND Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03842189/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03842189/SAP_001.pdf